CLINICAL TRIAL: NCT05290103
Title: Promoting Early Adolescent Non-smoking With a Game Intervention Supporting Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Johanna Nyman, Doctoral candidate, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEANS2022
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Self Efficacy; Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game intervention (Experimental): Participants in this arm will receive the game intervention including 15-30 minutes of digital health game playing at school and 2 weeks of free usage of the game during free time and a 30-minute debriefing session with a researcher.
  Interventions: Behavioral: Game intervention
- No intervention (No Intervention): The participants in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: Game intervention — Game intervention consists of 15-30 minutes digital health game playing at school and 2 weeks free usage of the digital health game during free time. In addition, after the 2 weeks period of game playing, 30-minute debriefing sessions with a research are held.
  The digital health game includes visualized elements with sound effects that aim at increasing understanding about the consequences of tobacco product use and supporting refusal skills. The health game includes different mini-games and also textual information.
  The debriefing sessions with a researcher include small group and group discussions about the themes presented in the game. A researcher leads and teachers facilitate the discussions. The debriefing sessions aim to connect the game experience with daily life situations.
  Arms: Game intervention

SUMMARY:
This intervention study evaluates the effectiveness of a digital game intervention supporting smoking refusal self-efficacy among early adolescents (10-13 y). The participants are randomly allocated to two groups: the experimental group that receives the digital game intervention, and the control group that receives no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Goes to school at 4th, 5th, or 6th grade
* Sufficient skills in Finnish or Swedish

Exclusion Criteria:

-

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 781 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Change in smoking refusal self-efficacy | At baseline, at 2 weeks, and at 3 months
  Assessed with a smoking refusal self-efficacy scale (scores 6-24; higher scores indicate stronger smoking refusal self-efficacy).

SECONDARY OUTCOMES:
Change in sources of refusal self-efficacy related to tobacco use | At baseline, at 2 weeks, and at 3 months
  Subscales for cigarette use (7 items) and snus use (7 items). Both are assessed with a 4-point Likert-scale questionnaire.
Change in motivation to decline tobacco use in the future | At baseline, at 2 weeks, and at 3 months
  Subscales for cigarette use and snus use. Both are assessed with a 4-point Likert-scale questionnaire (scores 1-4, lower scores indicate stonger motivation to decline tobacco use in future).

CONTACTS AND LOCATIONS:
Locations (1):
- Primary schools (n=15), Nine Cities, Finland

IPD SHARING:
Plan to Share IPD: No